CLINICAL TRIAL: NCT07383181
Title: The Effect of Standing and Squatting Positions During the First Stage of Labor on Birth Process, Birth Comfort, and Perceived Traumatic Birth Experience Among Multiparous Women
Brief Title: Standing vs. Squatting Positions During Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Nilgun Avci, Biruni University, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Standing vs. Squatting Positio
Record Dates: First submitted 2026-01-14; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Labor Position and Maternal Birth Experience

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standing Position Group (Experimental): Participants assigned to this group followed a standing position-based labor management approach during the first stage of labor.
  Interventions: Behavioral: Standing Position During Labor
- Squatting Position Group (Experimental): Participants assigned to this group followed a squatting position-based labor management approach during the first stage of labor.
  Interventions: Behavioral: Squatting Position During Labor

INTERVENTIONS:
Behavioral: Standing Position During Labor — Women were encouraged to remain standing or to walk during contraction-related pain episodes throughout the first stage of labor under midwife supervision.
  Arms: Standing Position Group
Behavioral: Squatting Position During Labor — Women were encouraged to assume the squatting position during contractions during the first stage of labor, supported by a birthing ball or bed rails according to preference.
  Arms: Squatting Position Group

SUMMARY:
Background: Maternal position during labor is a key non-pharmacological strategy that supports physiological birth and women's active participation in the childbirth process. Although upright positions have been associated with favorable labor outcomes compared with supine positions, evidence directly comparing different upright positions-particularly in relation to maternal birth experience and perceived traumatic birth-remains limited.

Objective: This study aimed to compare the effects of standing and squatting positions during the first stage of labor on the birth process, birth comfort, pain intensity, and perceived traumatic birth experience among multiparous women.

Methods: This study was conducted using a comparative interventional design. A total of 82 multiparous women were included and allocated to either the standing group (n=41) or the squatting group (n=41) during labor. Data were collected using a personal information form, the Visual Analog Scale (VAS) for pain, the Labor Comfort Scale, and the Traumatic Birth Perception Scale. Outcomes were assessed during labor and within the first two hours postpartum. Statistical analyses included comparative and correlation analyses.

ELIGIBILITY:
Inclusion Criteria:

* Multiparous women aged ≥18 years
* Gestational age between 38 and 42 weeks
* Singleton pregnancy with cephalic presentation
* Cervical dilatation ≥4 cm at admission
* Low-risk pregnancy
* Willingness to participate and provide written informed consent

Exclusion Criteria:

* Multiple pregnancy
* Presentation anomalies
* High-risk pregnancy (e.g., preeclampsia, gestational diabetes, placenta-related complications)
* Fetal distress or known fetal anomalies
* Any medical or obstetric condition requiring restricted mobility during labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Total Labor Duration | From active labor onset (cervical dilatation ≥4 cm) to delivery
  Total duration of labor measured in hours.
Birth Duration | From the active phase of labor to birth
  Duration of the birth process measured in minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Nilgün Avcı, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No